CLINICAL TRIAL: NCT05444673
Title: Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Brief Title: A Prospective, Single-arm Clinical Study of Pabrolizumab in Combination With Cisplatin + 5-FU for the Neoadjuvant Treatment of Unresectable, Advanced Squamous Carcinoma of the Temporal Bone Single-arm Clinical Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-KY-068
Record Dates: First submitted 2022-06-26; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Temporal Bone Squamous Cell Carcinoma
MeSH Terms: interventions — Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Paprizumab combined with cisplatin and 5-FU (Experimental): Patients received four cycles of paprizumab (200mg iv, 21-day cycle) in combination with 5-fu (500mg/m2 iv) plus cisplatin (80mg/m2 iv, 21-day cycle). Reassessment after completion of neoadjuvant chemotherapy was performed in operable patients.
  Interventions: Drug: Paprizumab combined with cisplatin and 5-FU

INTERVENTIONS:
Drug: Paprizumab combined with cisplatin and 5-FU — Patients with advanced temporal bone cancer were treated with pabulizumab combined with cisplatin and 5-FU

SUMMARY:
Temporal bone cancer accounts for 0.2% of head and neck cancers. Advanced temporal bone cancer often involves structures such as apices, internal carotid artery canals, and dura mater, and negative margins cannot be obtained during surgery. The recurrence rate after surgery is as high as 70%, and the 2-year survival rate is only 11%. Crestor, or paprolizumab, is a monoclonal antibody to PD1 that blocks the interaction between PD1 and the dura mater. The NCCN guidelines recommend that paprolizumab be used in combination with platinum-based anti-tumor agents. The NCCN guidelines recommend pablizumab in combination with platinum and 5-FU for the first-line treatment of recurrent, unresectable head and neck squamous carcinoma, but this regimen is not recommended for the treatment of recurrent, unresectable head and neck squamous carcinoma. This study is intended to investigate the use of pablizumab in combination with platinum and 5-FU for the first-line treatment of recurrent unresectable squamous head and neck cancer. This study investigates the effectiveness of pablizumab in combination with cisplatin and 5-FU for the adjuvant treatment of recurrent, unresectable temporal bone cancer. temporal bone cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced temporal bone carcinoma evaluated by an otolaryngologist as non-R0 resectable; CPS score > 20.
2. Patients who had undergone surgery, chemotherapy, radiotherapy, etc.
3. Patients with T4 advanced temporal bone cancer, Patients with nasopharyngeal carcinoma after radiotherapy
4. Hematology, biochemistry, and organ function:

   * Hemoglobin ≥100 g/L (can be maintained or exceeded by transfusion);
   * Neutrophil absolute count ≥2.0×109/L;
   * Platelet count ≥100×109/L;
   * Total bilirubin ≤1.5 times the upper limit of normal;
   * Alt and ASPARTate aminotransferase ≤2.5 times the upper limit of normal value;
   * Creatinine ≤1.25 times the upper limit of normal; The creatinine clearance rate was ≥60mL/min.
   * Women of childbearing age (18-49 years) must exclude pregnancy.
5. General admission criteria:

   * Obtain informed consent signed by the patient or his legal representative;
   * Good patient compliance;
   * Medications can be taken orally;
   * Male or female aged ≥18 years and < 75 years;
   * ECOG behavior status score 0-1, life expectancy > 12 weeks;
   * Both men and women of reproductive age agreed to use a reliable method of contraception before entering the trial, during the study, and up to 8 weeks after stopping the drug.

Exclusion Criteria:

Patients who had cancer other than temporal bone cancer during the five years before the initiation of treatment in this study were excluded from: fully cured with surgery and disease-free survival of at least 5 years; carcinoma in situ of the cervix; cured basal cell carcinoma; bladder epithelial neoplasms (including Ta and Tis);

* Known allergy to carboplatin, 5-FU, or any of the ingredients in this product;
* Confirmed or suspected active immune disease. The following conditions can be included: the absence of a specific external stimulus will not develop; Systemic treatment is not required.
* systemic use of steroid hormones (> 10mg/ day equivalent of prednisone) or immunosuppressants within 14 days before first administration. Aerosolized inhalation or topical administration of steroid steroids may be used in the absence of active immune disease.
* Previous interstitial lung disease, drug-induced interstitial disease, radiation pneumonia requiring hormone therapy, or any clinically proven active interstitial lung disease;
* Any unstable systemic disease, including: Active infection, uncontrolled hypertension, unstable angina, the onset of angina within the last 3 months, congestive heart failure (≥ New York Heart Association [NYHA] Class II), myocardial infarction (6 months before enrollment), severe arrhythmia requiring medication, liver, kidney, or metabolic disease;
* Known human immunodeficiency virus (HIV) infection, active hepatitis B or C;
* Patients with mixed small cell lung cancer components;
* Pregnant or lactating women;
* A clear history of neurological or psychiatric disorders, including epilepsy or dementia;
* Conditions deemed unsuitable for inclusion by other researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
The resectability rate of pablizumab in combination with cisplatin and 5-FU for unresectable temporal bone squamous carcinoma as neoadjuvant therapy | up to three months
  Resectability rate of tumors

CONTACTS AND LOCATIONS:
Overall Officials: Suijun CHEN, doctor, Study Director — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No